CLINICAL TRIAL: NCT04559503
Title: The Effect of Progressive Relaxation Exercises on Dyspnea and Anxiety Levels in Individuals With COPD
Brief Title: Progressive Relaxation Exercises in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Züleyha Kılıç, Assistant Professor, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OHU-zuleyha
Record Dates: First submitted 2020-09-13; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Anxiety; Dyspnea
MeSH Terms: conditions — Anxiety Disorders; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): Progressive relaxation exercises were applied once a day for four weeks in the intervention group in addition to the standard treatments. The patients were called 3 times each week on the telephone, and it was monitored whether they continued to do the exercises.
  Interventions: Other: Progressive relaxation exercises
- Control group (No Intervention): The control group received standard treatment.

INTERVENTIONS:
Other: Progressive relaxation exercises — Progressive relaxation exercises are those involving the voluntary, regular and consecutive relaxation of the muscles until there is relaxation all over the body. PMR are consisted of taking a deep breath and then tensing and relaxing muscles in both hands and arms, shoulders, chest, abdomen, hips, legs, feet, and face regions. The training was given in line with the CD that was prepared by the Turkish Psychologists Association as three-part relaxation exercises. The first part of the CD contains the definition, purpose and applications to consider when doing the exercises and a definition of 10-minute deep relaxation. In the second 30-minute section, relaxation exercises are explained accompanied by the sound of streams and oral instructions. The last section, which consists of 30 minutes, contains only relaxation music without instructions.
  Arms: İntervention Group

SUMMARY:
Background: This study aimed to determine the effect of progressive relaxation exercises (PMR) on dyspnea and anxiety level in individuals with COPD Methods: The study was conducted in the pretest-posttest randomized-controlled trial and completed with 44 COPD individuals, 22 interventions and 22 controls. PMR were applied once a day for four weeks in the intervention group in addition to the standard treatments. The control group received standard treatment.

DETAILED DESCRIPTION:
Background: This study aimed to determine the effect of progressive relaxation exercises (PMR) on dyspnea and anxiety level in individuals with COPD Methods: The study was conducted in the pretest-posttest randomized-controlled trial and completed with 44 COPD individuals, 22 interventions and 22 controls. PMR were applied once a day for four weeks in the intervention group in addition to the standard treatments. The control group received standard treatment. For data collection Questionnaire Forms, Patient Follow-Up Schedules, Modified Borg Scale (MBS), Modified British Medical Research Council Dyspnea Scale (mMRC), COPD Assessment Test (CAT), and Beck Anxiety Scale were used.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD,
* Must be able to competence to answer the questionnaire questions,
* Must be able to communicate verbally,
* Over 18 years of age,
* To have 2nd or 3rd grade COPD according to the GOLD Guide Staging System,
* To have 2 or more severe dyspnea according to the mMRC Dyspnea Scale,
* No medication changes have been made in the last three months,
* Not having received pulmonary rehabilitation in the last 6 months,

Exclusion Criteria:

* To have severe psychological disorders,
* To have non-COPD pulmonary diseases,
* To have cancer,
* To have renal failure,
* To have thyroid dysfunction,
* To have liver dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Modified Borg Scale | change from baseline score at the end of four weeks
  The Modified Borg Scale was developed by Borg in 1970 to measure the effort that is spent during physical exercise. It is a scale that is often used to assess the exertion dyspnea severity and resting dyspnea severity. There are 10 items that define the severity of the dyspnea according to their degrees. The scoring is made between 0 (none) and 10 (very severe)
Modified British Medical Research Council Dyspnea Scale | change from baseline score at the end of four weeks
  Fletcher et al. developed the mMRC Dyspnea Scale in 1940s when he worked on the respiratory problems of the coal workers. Then, the British Medical Research Board developed this scale more, and used to monitor the natural course of the disease. There are 5 grade (grade 0 to grade 4) that define the description of breathlessness on various physical activities, which cause dyspnea sense.
  Grade 0: breathless with strenuous exercise; Grade 1: short of breath when hurrying on level ground or walking up a slight hill; Grade 2: walked slower than people of the same age on level ground, and experienced breathlessness or the need to stop to breathe when walking on level ground at their own pace; Grade 3: stop to breathe after walking about 100 yards, or after a few minutes on level ground; and Grade 4: too breathless to leave the house, or breathless when dressing / undressing.
COPD Assessment Test | change from baseline score at the end of four weeks
  It was developed by Jones et al. in 2009. The Turkish reliability and validity of it was conducted in 2012 by Yorgancıoğlu et al. (2012). It is an easy, 8-item, and short scale that clinically measures the effects of COPD and deterioration in health conditions. The lowest score that can be received from the scale is 0, and the highest score is 40.
Beck Anxiety Scale | change from baseline score at the end of four weeks
  This scale, which can distinguish anxiety from depression, was developed by Beck et al. (1988). The validity and reliability studies of the scale were conducted for Turkey by Ulusoy et al. in 1998. The scale measures the frequency of the anxiety symptoms of the individuals with self-evaluation. It is a 4-Point Likert scale, and consists of 21 items. The scores range between 0 and 63. According to the scores received from the scale, the anxiety levels of patients are assessed as 0-7 points: minimal, 8-15 points: mild, 16-25 points moderate, 26 and above points: severe anxiety level.
Patient Follow-Up Schedule | change from baseline score at the end of four weeks
  The Patient Follow-Up Schedule is the form in which the first follow-up (the first interview), the second follow-up (the second interview after 4 weeks), the results of the respiratory function, and the emergency admission status of the patients were recorded by the researcher.

IPD SHARING:
Plan to Share IPD: No